CLINICAL TRIAL: NCT06468605
Title: A Phase 1 Open-Label Study to Evaluate the Safety, Tolerability and Efficacy of JCXH-211 (SElf-Replicating RNA IL-12) Intratumoral Injection in Patients With Recurrent or Progressive High-Grade Glioma
Brief Title: Safety, Tolerability and Efficacy of JCXH-211 in Patients With Recurrent or Progressive High-Grade Glioma
Acronym: SERIL
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Immorna, the funder withdrew the funds to run this study
Sponsor: Duke University (Other)
Responsible Party: Principal Investigator, Mustafa Khasraw, MBChB, MD, FRCP, FRACP, Professor of Neurosurgery, Duke University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00112350
Record Dates: First submitted 2024-06-15; First posted 2024-06-21 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Recurrent or Progressive High-grade Glioma
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JCXH-211 (Experimental): Open label single arm infusion of a single dose of JCXH-211, a self-replicating RNA (srRNA)-based human IL-12, administered intratumorally via convection-enhanced delivery (CED).
  Interventions: Biological: JCXH-211

INTERVENTIONS:
Biological: JCXH-211 — JCXH-211 is a lipid nanoparticle (LNP) encapsulated srRNA, encoding the human IL-12 protein.

SUMMARY:
This is a phase 1 open label study to establish the safety, tolerability, maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D), and preliminary efficacy of a single dose of JCXH-211. The study agent JCXH-211, is a self-replicating RNA (srRNA)-based human IL-12, administered intratumorally via convection-enhanced delivery (CED) to patients with recurrent or progressive high-grade glioma. Primary objective is to determine MTD or RP2D for a single dose on the study drug. Secondary outcomes include overall survival (OS) and progression-free survival (PFS) as assessed by modified mRANO 2.0.

DETAILED DESCRIPTION:
This is a Phase 1 open label study designed to assess the safety, tolerability, and MTD or RP2D of the study drug, JCXH-211 as administered by CED in patients with recurrent or progressive high-grade glioma based on radiographic findings including patients with recurrent IDH-wildtype GBM or recurrent IDH-mutated astrocytoma, who have progressed after receiving standard-of-care therapy.

A stereotactic biopsy will be performed prior to administration of the study drug to confirm viable tumor and a catheter will be implanted into the appropriate site which will be confirmed by Computed Tomography (CT) scan post-operatively. A continuous intratumoral infusion of JCXH-211 at the assigned dose level will be administered as in patient. An Ommaya reservoir will also be placed in the lateral ventricle at time of surgery to remove intracranial pressure by removing CSF and collect sample for exploratory analyses.

Patients will be followed up in clinic at 1 week and 2 weeks for adverse events (AEs),and subsequently for AEs and radiographic monitoring at 4 weeks, 8 weeks, and every 8 weeks thereafter until 48 weeks or disease progression, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old at the time of entry into the study
2. Recurrent or progressive high-grade glioma (Note: A frozen section diagnosis of recurrent glioma is necessary prior to placement of Ommaya reservoir and infusion catheter.) This includes:

   i. subjects with recurrent IDH wild-type GBM, who have recurred or progressed after prior treatment with radiation and TMZ (prior TMZ is mandated if known methylated MGMT promoter), and ii. subjects with recurrent IDH-mutated astrocytoma who have recurred after receiving standard therapy including radiation and chemotherapy, and either TMZ, lomustine or PCV [procarbazine, CCNU (lomustine) and vincristine].

   Note: Patients should be able to undergo tumor resection, regardless of glioma type.
3. Enhancing tumor volume of ≥ 10 mm x 1 mm amenable to CED catheter insertion per treating neurosurgeon
4. Karnofsky Performance Status (KPS) > 70%
5. Adequate organ function within 7 days prior to first administration of JCXH-211

   1. Platelets ≥ 100,000 per micro liter unsupported is necessary for eligibility on the study; however, because of risks of intracranial hemorrhage with catheter placement, platelet count ≥ 125,000 per micro liter is required for the patient to undergo biopsy and catheter insertion, which can be attained with the help of platelet transfusion.
   2. Hemoglobin ≥ 9 gm/dL
   3. Absolute neutrophil count (ANC) ≥ 1000 per micro liter
   4. Creatinine < 1.5 x upper limit of normal (ULN)
   5. Total bilirubin < 1.5 x ULN (Exception: Participant has known or suspected Gilbert's Syndrome for which additional lab testing of direct and/or indirect bilirubin supports this diagnosis. In these instances, a total bilirubin of ≤ 3.0 x ULN is acceptable.)
   6. AST/ALT < 2.5 x ULN
6. Prothrombin and Partial Thromboplastin Times ≤ 1.2 x normal prior to biopsy. Patients with prior history of thrombosis/embolism are allowed to be on anticoagulation, understanding that anticoagulation will be held in the perioperative period per the neurosurgical team's recommendations. Low molecular weight heparin (LMWH) is preferred. If a patient is on warfarin, the international normalized ratio (INR) is to be obtained and value should be below 2.0 prior to biopsy.
7. Able to undergo MRI of brain with and without contrast
8. If the patient is a sexually active female of childbearing potential whose partner is male, or if the patient is a sexually active male whose partner is a female of childbearing potential, the patient must use appropriate contraceptive measures for the duration of the treatment and for 6 months afterwards. Female patients of childbearing potential must have a negative serum pregnancy test at the time of screening and within 48 hours of starting the infusion of the study drug.
9. Signed informed consent approved by the IRB

Exclusion Criteria:

1. Prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
2. Patients who are pregnant or breastfeeding
3. Patients with contrast-enhancing tumor crossing the midline, multifocal tumor, infratentorial tumor, extensive tumor dissemination (subependymal or leptomeningeal), or in unsafe brain regions per the opinion of the treating neurosurgeon.
4. Patients with worsening neurologic deficits, clinically significant increased intracranial pressure (e.g., impending herniation), uncontrolled seizures, or requirement for immediate palliative treatment
5. Patients on > 2 mg per day of dexamethasone within the 1 week prior to admission for the infusion of the study drug. Please note: If a patient experiences adverse symptoms related to vasogenic edema causing significant symptoms after signing informed consent, additional steroids can be administered as indicated, but patient will be replaced for the purposes of PK analyses only (i.e., they will remain evaluable for safety/toxicity endpoints).
6. Patients who have not received standard of care treatments, including standard radiation and temozolomide, prior to participation in this trial (Please note: For patients under 65 years old, standard radiation therapy is typically at least 59 Gy in 30 fractions over 6 weeks. For patients 65 years or older, standard RT is often reduced to a minimum 40 Gy in 15 fractions over 3 weeks.)

   1. If the MGMT promoter in their tumor is known to be unmethylated, patients are not mandated to have received chemotherapy prior to participating in this trial.
   2. If the MGMT promoter in their tumor is known to be methylated or the MGMT promoter methylation status is unknown at time of screening, patients must have received at least one chemotherapy regimen prior to participating in this trial.
7. Less than 12 weeks from radiation therapy, unless progressive disease outside of the radiation field or 2 progressive scans at least 4 weeks apart or histopathologic confirmation of recurrent tumor.
8. Treated with immunotherapeutic agents within 4 weeks, alkylating agents within 4 weeks, nitrosoureas within 6 weeks, or non-alkylating chemotherapy within 2 weeks before enrolment, unless the patient has recovered from the expected toxic effects of such therapy.
9. Treated with antiangiogenic agents (i.e., bevacizumab) within 4 weeks before biopsy.
10. Patients may not have received treatment with tumor treating fields (e.g., Optune®) ≤ 1 week prior to starting the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
MTD or RP2D | Day 1 of treatment until 28 days post first infusion
  Determine Minimum Tolerated Dose (MTD) or Recommended Phase 2 Dose (RP2D) of JCXH-211 in patients with recurrent or progressive high-grade glioma

SECONDARY OUTCOMES:
Overall Survival | 5 years
  Day 1 of treatment until death to calculate Median overall survival by the Kaplan-Meier method.
Progression Free Survival | 5 years
  Day 1 of treatment until first documentation of disease progression as assessed by modified RANO 2.0 criteria or death to calculate Median progression free survival by the Kaplan-Meier method.

IPD SHARING:
Plan to Share IPD: No